CLINICAL TRIAL: NCT04564391
Title: Molke Oder Casein - Leberfettreduktion Und Stoffwechselverbesserung Durch Schnelle vs. Langsame Proteine (Whey or Casein - Liver Fat Reduction and Metabolic Improvement by Fast vs. Slow Proteins)
Brief Title: Whey or Casein - Liver Fat Reduction and Metabolic Improvement by Fast vs. Slow Proteins
Acronym: MOCA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Technische Universität Berlin (Other); University Hospital Tuebingen (Other); German Institute of Human Nutrition (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Andreas F. H. Pfeiffer, Head Dept. Endocrinology, Diabetes and Nutrition, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MOCA
Record Dates: First submitted 2020-07-21; First posted 2020-09-25 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Type2 Diabetes; NAFLD
Keywords: NAFLD; type 2 diabetes; whey protein; casein; second meal effect; pea protein
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: parallel-designed randomised controlled trial
Who Masked: Participant
Masking Description: For the preliminary meal tests all drinks and food supplements are provided in neutral bottles and cannot be identified by visual appearance, taste, texture or odour. Masking applied to participants, care providers, investigators and outcomes assessors.
  For the interventional study provided drinks and food supplements were masked best possible for the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Whey protein group, 60g/day (Active Comparator): Three weeks, daily supplementation with 60 g of whey protein
  Interventions: Dietary Supplement: protein supplement
- Casein protein group, 60 g/day (Active Comparator): Three weeks, daily supplementation with 60 g of casein protein
  Interventions: Dietary Supplement: protein supplement
- pea protein group, 60g/day (Active Comparator): Three weeks, daily supplementation with 60 g of pea protein
  Interventions: Dietary Supplement: protein supplement
- placebo arm (Placebo Comparator): Three weeks, daily supplementation with placebo
  Interventions: Dietary Supplement: placebo supplement

INTERVENTIONS:
Dietary Supplement: protein supplement — protein supplement, daily 60 g of protein, 3 weeks of intervention; blinded to patients
  Arms: Casein protein group, 60 g/day; Whey protein group, 60g/day; pea protein group, 60g/day
Dietary Supplement: placebo supplement — Placebo supplement, daily intake of placebo, 3 weeks of intervention; blinded to patients
  Arms: placebo arm

SUMMARY:
High-protein diets have been recently demonstrated to effectively reduce insulin resistance, derangements of the lipid profile and liver fat content in subjects with moderately and severely impaired glucose metabolism and non-alcoholic fatty liver disease (LeguAN, LEMBAS, DiNA-P, DiNA-D). The effects can be attributed to prolonged insulin secretion and improved second meal effect, higher energy expenditure by urea synthesis, suppression of glucagon or other mechanisms. Up to now, it is unclear, if proteins with slower or faster digestibility lead to differential results in these study designs. The proposed study will elucidate this question. The Investigators hypothesize, that slowly-digestible proteins induce a prolonged insulin plateau supporting the second-meal effect. The investigators also assume, that these dietary proteins lead to a markedly stronger short-term secretion of glucagon followed by desensitisation of this hormone release. Fast-digestible proteins, on the other hand, will presumably induce a smaller second-meal effect and do not inhibit a second rise of glucagon in a consecutive meal.

The investigators intend to study the effects of a 3-weeks high-protein diet in 80 subjects with NAFLD and T2DM on liver fat content (MR spectroscopy) and glucose metabolism. The investigators expect different results for slow protein (casein) and fast protein (whey), thus comparing both protein species. The two major clinical visits before and after the intervention period will include MRI spectroscopy, fasting blood sampling for later analysis, full anthropometric assessment, a mixed meal tolerance test and a set of behavioral tests, investigating decision making processes. In order to characterize the postprandial profiles (e.g. insulin, glucagon, amino acids) of the varying protein sources, preliminary meal tests are performed in overweight subjects with and without T2DM.

DETAILED DESCRIPTION:
High-protein diets have been recently demonstrated to effectively reduce insulin resistance, derangements of the lipid profile and liver fat content in subjects with moderately and severely impaired glucose metabolism and non-alcoholic fatty liver disease (LeguAN, LEMBAS, DiNA-P, DiNA-D). The effects can be attributed to prolonged insulin secretion and improved second meal effect, higher energy expenditure by urea synthesis, suppression of glucagon or other mechanisms. Up to now, it is unclear, if proteins with slower or faster digestibility lead to differential results in these study designs. The proposed study will elucidate this question. The investigators hypothesize, that slowly-digestible proteins induce a prolonged insulin plateau supporting the second-meal effect. They also assume, that these dietary proteins lead to a markedly stronger short-term secretion of glucagon followed by desensitisation of this hormone release. Fast-digestible proteins, on the other hand, will presumably induce a smaller second-meal effect and do not inhibit a second rise of glucagon in a consecutive meal.

The investigators intend to study the effects of a 3-weeks high-protein diet in 80 subjects with NAFLD and T2DM on liver fat content (MR spectroscopy) and glucose metabolism. The investigators expect different results for slow protein (casein) and fast protein (whey), thus comparing both protein species. The two major clinical visits before and after the intervention period will include MRI spectroscopy, fasting blood sampling for later analysis, full anthropometric assessment, a mixed meal tolerance test and a set of behavioral tests to investigate decision making processes.

In order to characterize the postprandial hormonal and amino acid profiles (e.g. insulin, glucagon, amino acids) of the varying protein sources, preliminary meal tests are performed. The first tests assess the protein dose-finding in 20 participants, 10 with T2DM and 10 without. On each day of the dose-finding assessment pre-trial one of the following dosages is used in a single oral protein tolerance test (5 g, 10 g and 30 g of whey or casein each).The second tests assess whether 30 g mixes of whey and casein in variable proportions induce different hormonal profiles of glucagon and insulin in comparison with 30 g pea protein, served as drinks together with a standardized breakfast. Therefore, 20 subjects, 10 with Metabolic Syndrome and T2DM and 10 with Metabolic Syndrome without T2DM undergo seven separate investigation days. The third preliminary tests assess the role of the product matrix/consistency in 6 participants with overweight/obesity. Participants consume commercially available milk products each 30 g protein content (approx. 80% Casein) but with different product consistency on three separate investigation days. Subjects without prior diabetes diagnosis additionally undergo an initial oral glucose tolerance test (OGTT) to ensure healthy glucose levels.

All clinical assessments will be conducted in the Dept. Endocrinology, Diabetes and Nutrition, Charité, Campus Benjamin Franklin (Lead: Charité, A.F.H. Pfeiffer). Psychobehavioral tests (DIfE, Prof. Park), assessment of body fat distribution including liver fat (University Hospital Tuebingen, Dr. Machann) and measurements of amino acid levels throughout the meal tests (Technische Universität Berlin, Prof. Rohn) are secondary work packages.

ELIGIBILITY:
Subcohort 1 (n=46):

Inclusion Criteria:

* healthy glucose levels or T2DM
* 40-79 years
* overweight/obesity

Main Exclusion Criteria:

* type 1 diabetes, prediabetes
* currently receiving treatment with insulin
* lactose intolerance, or food intolerance/allergy to any of the study products
* severe endocrine, gastrointestinal, metabolic, cardiovascular, pulmonary, inflammatory or psychiatric disorder
* active or recent relevant cancer
* intake of glucocorticoids or other medication that influences glucose metabolism
* pregnancy, breastfeeding

Subcohort 2 (n=80):

Inclusion Criteria:

* T2DM
* with NAFLD
* 18-79 years

Main Exclusion Criteria:

* type 1 diabetes, prediabetes
* currently receiving treatment with insulin
* lactose intolerance, or food intolerance/allergy to any of the study products
* severe endocrine, gastrointestinal, metabolic, cardiovascular, pulmonary, inflammatory or psychiatric disorder
* active or recent relevant cancer
* intake of glucocorticoids or other medication that influences glucose metabolism
* pregnancy, breastfeeding
* claustrophobia

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-09-21 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Liver fat change after three weeks | 3 weeks
  absolute liver fat reduction after three weeks (MR spectroscopy)
change of 2-hours glucose levels in mixed meal test | 3 weeks
  change of 2-hours glucose levels in mixed meal test
change of glucagon concentration pg/ml (ELISA) in mixed-meal test | 3 weeks
  change of glucagon concentration (pg/ml) in mixed-meal test
change of insulin concentration (mIU/ml) in mixed-meal test | 3 weeks
  change of insulin concentration (mIU/ml) in mixed-meal test calculated as (disposition index)
change of dynamic insulin sensitivity in mixed-meal test | 3 weeks
  change of dynamic insulin sensitivity in mixed-meal test (Matsuda)
change of fasting insulin sensitivity in mixed-meal test | 3 weeks
  change of fasting insulin sensitivity in mixed-meal test (HOMA-IR)

SECONDARY OUTCOMES:
change of insulin secretion in consecutive mixed-meal test after an initial breakfast MMT | 3 weeks
  change of insulin secretion in consecutive mixed-meal test after an initial breakfast MMT
change of urea concentration in serum(mmol/l) | 2 weeks
  change of urea concentration in Serum (mmol/l)

OTHER OUTCOMES:
change in fasting amino acid concentration in blood | 3 weeks
  change in fasting amino acid concentrations determined by LC-MS in blood
change in uric Acid concentration in Serum (µmol/l) | 3 weeks
  change in uric Acid concentration in Serum (µmol/l)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas FH Pfeiffer, Prof. Dr., Study Director — Charité Universitätsmedizinh Berlin
Locations (1):
- Charité Campus Benjamin Franklin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang J, Schafer SM, Kabisch S, Csanalosi M, Schuppelius B, Kemper M, Markova M, Meyer NMT, Pivovarova-Ramich O, Keyhani-Nejad F, Rohn S, Pfeiffer AFH. Implication of sugar, protein and incretins in excessive glucagon secretion in type 2 diabetes after mixed meals. Clin Nutr. 2023 Apr;42(4):467-476. doi: 10.1016/j.clnu.2023.02.011. Epub 2023 Feb 21. PMID 36857956